CLINICAL TRIAL: NCT05774210
Title: Cost of Disease and Falls Among Individuals With Parkinson's Disease Living in Hong Kong:
Brief Title: Cost of Parkinson's Disease in Hong Kong
Acronym: Burden of PD
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Chinese University of Hong Kong (Other); The University of Hong Kong (Other)
Responsible Party: Sponsor
Other Study IDs: HMRF_SW_2023
Record Dates: First submitted 2023-03-07; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-02

CONDITIONS: Parkinson Disease
Keywords: Cost of illness; Falls; PD; Disease burden
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this study is to estimate the cost of disease and falls among people with Parkinson's disease in Hong Kong . There will be no intervention delivered to the participants.

The healthcare cost of 12 months will be recorded using self-report and and the Hospital Authority Clinical Management System.

DETAILED DESCRIPTION:
Objective: Estimate the cost of disease and falls among people with Parkinson's disease in Hong Kong.

Design: Prospective cost-of-illness analysis with one baseline assessment and two follow-up assessments after 6 and 12 months.

Participants: Community-dwelling participants with Parkinson's disease. Intervention: N/A. Outcome measures: Self-reported questionnaires and the Hospital Authority Clinical Management System will be used to inform the healthcare utilisation. We will also assess the number of falls, severity of Parkinson's disease, level of disability, balance, risk of falls, and quality of life. Predictors of cost include fall frequency, balance status, disease severity, level of disability, quality of life and disease duration.

Analysis: Cost-of-illness analysis will estimate the direct and indirect cost, using a prevalence-based approach, by converting physical units to monetary value based on unsubsidised charges for healthcare in Hong Kong published by the Hospital Authority for the year 2022. A multiple regression analysis will determine predictors influencing the overall cost. A two-way ANOVA will assess differences in healthcare costs among frequent, infrequent and non-fallers. Sensitivity analysis will include (1) tornado plots for studying the degree of impact of the cost variables on mean cost, (2) analysis after removing cost outliers and (3) varying the expenses on selected cost items by 25%.

ELIGIBILITY:
Inclusion Criteria:

Community-dwelling participants with a confirmed diagnosis of Parkinson's disease Reside in Hong Kong

Exclusion Criteria:

Patients who are bedridden or solely wheelchair users, Have atypical Parkinson's syndrome and Have other associated major illnesses, such as stroke.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Community-dwelling patients with a confirmed diagnosis of Parkinson's disease who attend the outpatient clinics of the Prince Wales Hospital, Shatin and Queen Mary Hospital, Pok Fu Lam will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Client Service Receipt Inventory - RAre disease (CSRI-Ra) | Change score after 6 months and 12 months
  The CSRI is a widely used measure for recording cost-related data. The measure covers five key sections including background information, household and carer support, healthcare service and resource utilization, community support and education and employment. The CSRI-Ra is cross-culturally validated for Hong Kong Population (reference added to appendix 3a). The Chinese version of the self-reported CSRI-Ra both the patient version and carers version will be used in this study. The cost data will be captured across 6 months retrospective period. The background section 1 will be completed during the baseline assessment (T1) and sections 2 onwards will be completed during T2 and repeated during T3 assessment timelines.

SECONDARY OUTCOMES:
Number of falls | Change score after 6 months and 12 months
  We define a fall as any rapid and uncontrolled change from a sitting or upright position to a reclining position or the ground. Based on the number of falls, we define frequent fallers as those who have fallen five or more times, infrequent fallers as those with four or fewer falls, and non-fallers as those with no falls over 12 months
The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | Change score after 6 months and 12 months
  MDS-UPDRS is a measure of Parkinson's disease severity. The scale is scored from 0 to 199, with 0 indicating no disability and 199 indicating maximal disability due to disease. Severity is scored across five segments, including (i) mental, behavior and mood, (ii) activities of daily living (ADL), (iii) motor examination, (iv) the modified Hoehn and Yahr Scale, and (v) the Schwab and England ADL scale.
Hoehn and Yahr Scale | Change score after 6 months and 12 months
  The Hoehn and Yahr Scale is a measure for the level of disability due to Parkinson's disease. The scale classifies the patient from Stage 0 (no disease signs) to Stage 5 (bedridden or solely mobile by wheelchair).
Falls Efficacy Scale-International (FES-I) | Change score after 6 months and 12 months
  The FES-I is a self-reported measure for assessing the fear of falls among community-dwelling older adults. The scale includes 16 items, scored between 1 and 4. The scale has a minimum score of 16, which indicates no concerns regarding falls, and a maximum score of 64, indicating maximal concern regarding falls. The FES-I is a valid measure for estimating the fall risk among people with Parkinson's disease
Activities-Specific Balance Confidence Scale (ABC) | Change score after 6 months and 12 months
  The ABC is a non-disease-specific, self-reported measure of balance confidence. The scale includes 16 items, each rated between 0%, indicating no confidence, and 100%, indicating complete confidence regarding the activity in question. Higher scores indicate better balance performance. The ABC is both reliable and valid for the assessment of balance in people with Parkinson's disease
Short-Form Health Survey (SF-36) | Change score after 6 months and 12 months
  Quality of life will be measured using the SF-36. The scale has eight domains, each scored between 0 and 100, with 0 interpreted as worst health and 100 as the best health status.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley J Winser, PhD, Principal Investigator — The Hong Kong Polytechnic University